CLINICAL TRIAL: NCT07168642
Title: A Type I Hybrid Effectiveness-Implementation Trial of Mothering From the Inside Out (MIO)
Brief Title: A Type I Hybrid Effectiveness-Implementation Trial of MIO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baystate Medical Center (Other)
Collaborators: Behavioral Health Network (Unknown); Spectrum Health Systems (Unknown)
Responsible Party: Principal Investigator, Elizabeth Peacock-Chambers, MD, Associate Professor of Pediatrics, Division Chief of Health and Behavior, Baystate Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BH-25-127
Record Dates: First submitted 2025-08-13; First posted 2025-09-11 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Substance Use Disorder
Keywords: substance use disorder; parenting; parenting intervention; Mothering from the Inside Out; MIO; SUD treatment
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Mothering from the Inside Out (MIO) + treatment as usual (TAU)
  Interventions: Behavioral: Mothering from the Inside Out
- Control (No Intervention): Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Mothering from the Inside Out — Mothering from the Inside Out (MIO) is an evidence-based individual psychotherapy designed to help caregivers in recovery build stronger relationships with their children. In MIO, caregivers are helped to build their ability to reflect on their own mental states and how they arose. Often, we find that the thoughts and feelings that drive caregiving behavior are actually triggered by early experiences of being cared for. MIO thus aims to provide a safe, therapeutic space where caregivers' internal experiences are taken seriously and clinicians are genuinely interested, curious, and collaborative. MIO also involves helping caregivers to reflect on the possible mental states underlying their children's behavior. We find that by providing some information about child development through an attachment lens, this can help parents see through their children's eyes and feel less stressed.
  Arms: Intervention

SUMMARY:
Mothers with substance use disorders face unprecedented stress in their roles as parents working to care for their children while maintaining healthy recovery. Mothering from the Inside Out (MIO) is the first attachment-based parenting intervention designed specifically for mothers in recovery from substance use disorders that has been shown to have benefit for both mother and child in multiple randomized controlled trials. This project will: (a) test the effectiveness of MIO among women in outpatient treatment under 'real-world' conditions, (b) evaluate implementation in different settings, and (c) assess key implementation factors to support optimal uptake and treatment in future dissemination studies; closing an important science-to-service gap for an underserved population in an effort to support maternal and child health simultaneously.

DETAILED DESCRIPTION:
Pregnancy and parenting can be life-changing motivators for women with substance use disorders (SUDs) to seek treatment. However, the rate of relapse and overdose for women with SUDs increases sharply after the birth of a child, such that mental health and drug-related deaths are a leading preventable cause of postpartum mortality. Heightened parental stress and lack of adequate parenting supports increase the risk of drug overdose. Mothers with SUDs are also more likely to exhibit maladaptive parenting behaviors associated with long-term developmental, behavioral, and emotional problems in their offspring. Despite the well-established interaction between parenting and SUDs during a critical period, SUD treatment does not systematically include targeted parenting support for mothers in recovery and their young children.

Mothering from the Inside Out (MIO) is an evidence-based, individual parenting intervention designed as an adjunct to outpatient SUD treatment that targets parental reflective functioning, i.e., the capacity to understand behavior, for oneself and one's child, in terms of underlying mental states. MIO has proven bigenerational efficacy in two randomized trials when delivered by researchers under tightly controlled research conditions. Mothers assigned to MIO demonstrated significantly improved parenting capacities and reduced substance use compared with those assigned to parental education.

Although MIO was efficacious when delivered by expert clinicians in highly organized research settings, there are challenges to exporting any evidence-based practice to dynamic real-world environments creating a science-to-service gap. As a first step in addressing these challenges, we successfully trained SUD and mental health counselors to deliver MIO with fidelity in community clinics. Yet, in the only community-based efficacy trial where MIO was delivered by SUD treatment counselors, MIO offered some advantages over parental education with respect to reduction in substance use and depressive symptoms, but MIO did not yield the same magnitude of improvement in parenting as it did in the first two randomized controlled trials.

Community-academic partnerships and governmental funding support in Massachusetts have since allowed our multi-disciplinary team to identify barriers to implementation and develop a practice-informed implementation strategy to mitigate these barriers. We are now poised to simultaneously test the clinical effectiveness of MIO and the utility of our implementation strategy in community-based clinical settings. With guidance from our two community partners, we are proposing a Hybrid Type II research project to test the effectiveness and implementation of MIO as an adjunct to treatment as usual (TAU). SUD counselors (n=16) and mothers enrolled in outpatient SUD treatment (n=200) caring for children ≤5 years of age will be recruited from four SUD treatment clinics operated by two community agencies in Massachusetts. These sites were selected by our community partners based on their generalizability and engagement with parents with SUDs. Mothers will be randomized in a 2:1 fashion to the receipt of either MIO+TAU or TAU to allow for dual examination of the implementation process as well as the MIO mechanism of change. Guided by established frameworks and our implementation conceptual model, we will use a mixed-methods approach to evaluate the relationship between key contextual determinants of MIO implementation. Our specific aims include the following:

Aim 1. Compare the effectiveness of MIO+TAU versus TAU alone. Hypotheses: Compared with mothers receiving TAU, mothers randomized to MIO+TAU will demonstrate a greater increase in parental reflective functioning and greater decrease in parenting stress (primary outcomes) at the end of treatment. They will also demonstrate greater improvement in quality of mother-child interactions and greater decreases in drug use and psychiatric distress (secondary outcomes) at 3-month follow-up.

Aim 2. Assess differences in agency- and clinic-level implementation processes with respect to a) completion of implementation activities, b) tailoring strategies, and c) implementation outcomes.

Hypothesis: Facilitated completion of pre-implementation activities at the agency- and clinic-level will predict greater reach, adoption, feasibility, and fidelity of MIO across four clinical units.

Aim 3. Identify key contextual determinants associated with successful MIO implementation and effectiveness, supported by integration of qualitative and quantitative data to guide large-scale dissemination.

Hypothesis 3a: Primary implementation outcomes (MIO fidelity and feasibility) will be determined by organizational climate, characteristics of individual counselors, and execution of the implementation process integrity.

Hypothesis 3b: The association between primary implementation outcomes (MIO fidelity and feasibility) and secondary effectiveness outcomes (quality of mother-child interactions, maternal drug use, and psychiatric distress) will be mediated by parental reflective functioning and parenting stress (primary effectiveness outcomes).

Moving evidence-based practices into routine care settings is a public health and NIDA priority. When completed, this project will allow us to address the critical gap between research and practice by providing data to support large-scale implementation of MIO in community settings.

ELIGIBILITY:
Client Subjects

Inclusion Criteria:

* Identifies as a woman
* English-speaking
* Age 18 years or older
* Enrolled in outpatient substance use treatment for a substance use disorder (by DSMV criteria) at one of the four target clinics operated by participating agencies
* Caring for at least one child between 0 and 60 months of age (either as guardian or working towards reunification with regular contact)

Exclusion Criteria:

* Have severe mental health problems (e.g., actively suicidal, homicidal, psychosis)
* Severely cognitively impaired
* Have psychiatric or substance-related symptoms requiring inpatient hospitalization or ambulatory detoxification
* Unable to speak English
* Have a potential target child who has a severe medical condition that limits their ability to interact with their mother (such as paralysis or severe weakness)

Children Subjects

Inclusion Criteria:

* Age 5 years or younger
* Are in their biological mother's custody OR are in custody of family with the goal of reunification with their biological mother and have permission from the child's legal guardian to participate in this study

Exclusion Criteria:

•In child welfare custody and goal is not reunification with biological mother

Counselor Subjects

Inclusion Criteria:

* Age 21 years or older
* Employed as an addiction counselor at one of the participating agencies in one of the target clinics
* Have a bachelor's degree or higher in psychology, social work, counseling, or a related field
* Have secure administrative approval for a 1-hour per biweekly commitment to supervision and 2-3 hours weekly for MIO delivery
* Do not intend to give notice and are not scheduled for medical or family leave during the study period
* Willing to have counseling and supervision sessions recorded
* Receive a mean score greater than 4 on the Clinical Reflective Functioning Scale
* Are deemed capable to manage the responsibilities of being a counselor in a randomized trial (deliver MIO promptly to participants, compliant with study procedures and assessments, willing to receive supervision) by their supervisors

Exclusion Criteria:

•None

Agency Staff Subjects

Inclusion Criteria:

* Employment at a participating agency for at least 3 months
* Willingness to complete questionnaires and participate in a confidential interview or focus group
* Fluency in English

Exclusion Criteria:

•None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Parents that identify as mothers
Enrollment: 200 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Parental Reflective Functioning | Baseline, post treatment (week 21)
  The Parent Development Interview (PDI) is a semi-structured clinical interview with 19 questions intended to examine parents' representations of their children, themselves as parents, and their relationships with their children. The PDI is coded using an 11-point reflective functioning rating scale (-1 to 9) where higher score indicates higher reflective capacity.
Parental Reflective Functioning | Baseline, post treatment (week 21)
  The Parental Reflective Functioning Questionnaire (PRFQ) is an 18-item questionnaire assessing caregiver's capacity to reflect upon his/her own internal mental experiences as well as those of the child. Uses a 7-point Likert scale with 1 being "Completely disagree," 4 being "Neutral," and 7 being "Completely agree." Items 11 and 18 are reverse coded. Minimum score is 18, max is 126. High scores on this scale indicate serious distortions in parental reflective functioning.
Parenting Stress | Baseline, during treatment (week 13), post treatment (week 21), follow-up (week 33)
  The Parenting Stress Index-Short Form (PSI-SF) is a 36-item questionnaire used to assess parenting stress on a 5-point Likert scale. It's a briefer version of the full Parenting Stress Index, designed to be more efficient for clinical and research settings. The PSI-SF measures three key areas: Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child, which together contribute to an overall measure of parenting stress, minimum score 36 and maximum 180. Scores at or above the 85th percentile on the Total Stress scale are considered to be borderline clinically significant.

SECONDARY OUTCOMES:
Quality of mother-child interaction | Baseline, follow-up (week 33)
  The Coding Interactive Behavior (CIB) is a global rating system for analyzing social interactions between two or more partners, in this case, mother and child (videotaped play session with recommended age-appropriate toys). The CIB consists of 33 items (18 relating to the parent, 8 to the child, 5 to the dyad, and 2 focusing on the lead-lag of the interaction) that are rated from 1 (minimal level of behavior) to 5 (maximum level of behavior). Minimum possible score is 33, maximum is 165. A higher score indicates a more positive and adaptive interactive behavior between parent and child.
Substance Use | Baseline, monthly during weeks 1-21, post treatment (week 21)
  Toxicology testing is a method to detect the presence of drugs or other chemicals in a person's urine. This testing is already being completed as a normal procedure by the SUD treatment agencies, and the results on study participants only are shared with the study team on a monthly basis.
Substance Use | Baseline, during treatment (week 13), post treatment (week 21), follow-up (week 33)
  The Timeline Followback (TLFB) is a method to assess recent drug use. It involves asking clients to retrospectively estimate their drug use 7 days to 2 years prior to the interview date. TLFB data can be scored in various ways to quantify different aspects of substance use - for this study, we are looking at whether participants have recent drug use or not.
Anxiety | Baseline, during treatment (week 13), post treatment (week 21)
  The General Anxiety Disorder-7 (GAD-7) is a 7-item screening tool used to assess the severity of generalized anxiety disorder. Each item is rated on a 0-3 scale, with higher scores indicating greater anxiety. Minimum score 0, maximum score 21.
Depression | Baseline, during treatment (week 13), post treatment (week 21)
  The Patient Health Questionnaire-9 (PHQ-9) is a self-administered tool used to screen for and assess the severity of depression. It consists of nine questions, each scored from 0 (not at all) to 3 (nearly every day), with a total possible score ranging from 0 to 27. Higher scores indicate more severe depression, and scores are categorized into ranges to suggest severity levels: minimal (0-4), mild (5-9), moderate (10-14), moderately severe (15-19), and severe (20-27).
MIO Fidelity | Intervention period weeks 4-21
  Mothering from the Inside Out - Treatment Fidelity Scales - Revised (MIO-TFS-R) is used to code MIO sessions in frequency and competence across 10 competencies with scores for each competency ranging from 0 to 3. Four of these competencies are MIO-specific, with higher scores on MIO items indicating greater fidelity to the MIO model. For both frequency and competence, the minimum possible overall score is 10 the maximum possible overall score is 30. The minimum score for MIO-specific items is 4, and the maximum is 12.
MIO Feasibility | After each MIO treatment (week 21 of each mother's participation period)
  Number of MIO sessions completed in a 16-week period
Organizational Culture | Years 1 & 5
  The Organizational Climate Measuring Tool (OCMT) is a standardized scale measuring agency culture. It uses a Likert-type scale of 10 points (1 = maximum disagreement; 10 = maximum agreement) to examine motivation, leadership, and management philosophy.
Organizational Attitudes | Years 1 & 5
  The Evidence-Based Practice Questionnaire (EBPQ) measures individuals' attitudes towards, knowledge of, and implementation of evidence-based practice, and the extent to which barriers may prevent greater uptake of evidence-based practice. The questionnaire contains 24 items scored on a seven-point Likert scale, with lower scores corresponding to poor attitude. There are 3 subscales: practice of evidence-based practice (6 items), attitude towards evidence-based practice (4 items), and knowledge/skills associated with evidence-based practice (14 items).

CONTACTS AND LOCATIONS:
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lowell AF, Peacock-Chambers E, Zayde A, DeCoste CL, McMahon TJ, Suchman NE. Mothering from the Inside Out: Addressing the Intersection of Addiction, Adversity, and Attachment with Evidence-Based Parenting Intervention. Curr Addict Rep. 2021;8(4):605-615. doi: 10.1007/s40429-021-00389-1. Epub 2021 Jul 15. PMID 34306964
- See also: Related Info — https://www.motheringfromtheinsideout.org/